CLINICAL TRIAL: NCT06892457
Title: PHArmacotherapy Assessed Using Neuroprobing With TransOsseal Magnetic Stimulation
Acronym: PHANTOMS
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 5958
Record Dates: First submitted 2025-03-21; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
Keywords: Brain Excitability; Anti-Seizure Medication; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: TMS-EEG — Evoked brain activity is measured with the help of TMS-EEG in epilepsy patients OFF and ON medication.

SUMMARY:
The goal of this observational study is to investigate how prescribed anti-seizure medications (ASMs) affect cortical excitability in adults with epilepsy. The main questions it aims to answer are:

1. Does the magnitude of transcranial magnetic stimulation (TMS)-evoked potentials (TEPs) measured with electroencephalography (EEG) change between OFF and ON medication states?
2. Do these changes in TEP amplitude persist over time? Researchers will compare each participant's measurements in the OFF state with those in the ON state to see if TEPs change following ASM (re)start.

Participants will undergo one TMS-EEG session scheduled around their prescribed ASM (re)start and one 1-6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18j) with epilepsy receiving a prescription for an anti-seizure medication for clinical reasons
* Written informed consent

Exclusion Criteria:

* Presence of any electrical implants (e.g. neurostimulator or drug delivery system) or any metallic implants anywhere in the head (excluding teeth)
* Increased intracranial pressure
* Uncontrolled psychiatric disorder
* Use of any kind of drug or alcohol, nicotine allowed
* For female participants: If pregnancy cannot be ruled out with sufficient certainty, a pregnancy test (urine) will be carried out before using TMS
* Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18j) with epilepsy receiving a prescription for an anti-seizure medication for clinical reasons.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Change in TEP magnitude | 1 day
  Whether the magnitude of measured TMS-evoked potentials (TEPs), measured as the line-length, is reduced between the OFF and ON ASM conditions.

SECONDARY OUTCOMES:
Persistence of TEP changes over time. | 1-6 months
  Number of participants with persistence of TEP changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Friedrichs-Maeder, MD, MSc., Principal Investigator — Bern University Hospital
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided